CLINICAL TRIAL: NCT07303478
Title: Comparison of Obturation Quality and Lateral Canal Fill (by Sealer): Ultrasonic-Activated Versus Non-Ultrasonic Conventional Irrigation Techniques in Root Canal Treatment - A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prime Foundation (Other)
Responsible Party: Principal Investigator, Syed Shahbaz Ali Shah, Doctor, Prime Foundation
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Prime Foundation
Record Dates: First submitted 2025-11-27; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Comparison Between Two Type of Irrigation Systems

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ULTRASONIC IRRIGITATION TECHNIQUE (Other)
  Interventions: Other: ULTRASONIC IRRIGATION TECHNIQUE
- NON-ULTRASONIC CONVENTIONAL IRRIGATION TECHNIQUE (Other)
  Interventions: Other: NON-ULTRASONIC CONVENTIONAL IRRIGATION TECHNIQUE

INTERVENTIONS:
Other: ULTRASONIC IRRIGATION TECHNIQUE — The utilization of theVAT-3 ultrasonic activator high frequency device (45KHz± 5kHz) [Refine] for the Ultrasonic Activated Irrigation group and same solution of 3% sodium hypochlorite and Tg Sealer will be used. Post-operative radiographs will be obtained to assess the obturation quality and lateral canal fill. A detailed radiographic proforma will be employed to evaluate the length, density, taper of the root canal filling, and lateral canal fill . Each of these components will be scored individually, and an overall Obturation Quality Score is calculated by summing these scores.
  Arms: ULTRASONIC IRRIGITATION TECHNIQUE
Other: NON-ULTRASONIC CONVENTIONAL IRRIGATION TECHNIQUE — The root canal treatment is then performed as per the assigned group, with conventional irrigation involving the use of syringes and 3% sodium hypochlorite solution and Tg Sealer for the Non-Ultrasonic Conventional Irrigation group.A detailed radiographic proforma will be employed to evaluate the length, density, taper of the root canal filling, and lateral canal fill . Each of these components will be scored individually, and an overall Obturation Quality Score is calculated by summing these scores.
  Arms: NON-ULTRASONIC CONVENTIONAL IRRIGATION TECHNIQUE

SUMMARY:
The main goal of clinical trail to compare obturation quality and lateral canal sealer fill between ultrasonic activated and conventional irrigation in root canal treatment.

HYPOTHESIS There is a difference in obturation quality and lateral canal fill between ultrasonic activated irrigation results as compared to conventional irrigation technique in root canal treatment.

Eligible patients will be recruited from the Endodontics Department at Peshawar Dental College who present with pain and sensitivity in mandibular teeth and are advised root canal treatment after clinical examination and X-ray. Patients will be screened according to inclusion and exclusion criteria and informed written consent will be taken. This will be a double-blinded study, and demographic and tooth-related information will be recorded.

Participants will be randomized into two groups using block randomization with a block size of six. The Non-Ultrasonic group will receive conventional irrigation using syringe, 3% sodium hypochlorite, and Tg sealer, while the Ultrasonic group will be irrigated using the VAT-3 ultrasonic activator with the same solution and sealer. Pre- and post-operative radiographs will be taken to evaluate obturation quality and lateral canal fill in terms of length, density, and taper using a standardized proforma.

ELIGIBILITY:
Inclusion Criteria:

* Both male and female
* Age group adults 18 to 70 years
* Patients presenting with pain and sensitivity in mandibular molars and advised root canal treatment after examination and x ray

Exclusion Criteria:

* Teeth with complex root canal anatomy that may complicate the obturation process
* Pregnancy
* Medically compromised patients including uncontrolled diabetes -cardiovascular disease immunodeficiency disorders bleeding disorders and -severe respiratory disease
* Patients who refused to participate in this study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
To compare obturation quality and lateral canal sealer fill between ultrasonic activated and conventional irrigation in root canal treatment | Immediate, after completion of procedure
  Obturation Quality and Lateral Canal Fill:- This will involve evaluating the length of the root canal filling in the main canals, assessing the homogeneity (density) of the obturation material, determining the taper of the root canal filling, and examining the sealer's penetration into lateral canals using postoperative radiographs. The radiographs will be reviewed independently by two senior endodontists. A scoring system will be applied, and each of the three parameters will be individually assessed.
  Lateral Canal:- A type of accessory canal located in the coronal or middle third of the root, usually extending horizontally from the main canal space.

CONTACTS AND LOCATIONS:
Locations (1):
- Peshawar Dental Collge, Peshawar, Khyber Pakhtoon Khawa(KPK)a, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after completion of results.
Access Criteria: Researchers studying similar primary outcomes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-04-30): https://cdn.clinicaltrials.gov/large-docs/78/NCT07303478/Prot_SAP_ICF_000.pdf